CLINICAL TRIAL: NCT02572193
Title: To Assess the Feasibility of Same Day Discharge Following a POEM Procedure
Acronym: POEM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015H1
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Achalasia
Keywords: achalasia; surgery
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active case (Experimental): POEM procedure
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — To determine the feasibility of same-day discharge following a POEM procedure

SUMMARY:
This is a study of an investigational surgical procedure for the treatment of achalasia the inability of smooth muscle to move food down the esophagus. A new procedure, called the POEM procedure (per oral endoscopic myotomy) has been developed for achalasia. This study is being performed to determine if patients can go home on the same day as their procedure.

DETAILED DESCRIPTION:
This is a study of an investigational surgical procedure for the treatment of achalasia the inability of smooth muscle to move food down the esophagus.

Standard care for participants includes Heller Myotomy, a laparoscopic procedure that includes cutting the muscle layers in the lower esophageal sphincter (LES) the valve at the bottom of your esophagus. A second procedure is then required to prevent reflux (acid entering the esophagus from the stomach) called fundoplication. Patients with the Heller myotomy will typically stay overnight in hospital. A new procedure, called the POEM procedure (per oral endoscopic myotomy) has been developed for achalasia. This procedure uses endoscopy and no incisions to cut one muscle layer. A fundoplication is not required with this method. This study treatment works by entering the surgical area through the mouth and then making an incision (cut) through the esophagus and placing flexible instruments along the outside of the esophagus and down to the LES through a tunnel. The instruments used in this procedure are standard endoscopic instruments that will be provided by one of the leading endoscopic instrument manufacturers, Olympus. The investigators have recently completed a small study showing this procedure is safe and feasible. One observation from this pilot study was that most patients had no pain and didn't need any pain medications. Due to this reason, the investigators think patient's may go home on the same day as their procedure.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet ALL of the following inclusion criteria:

* Candidate for a Heller myotomy
* Their age is ≥18 years and ≤80 years
* Able to give written consent

Exclusion Criteria:

Participants who meet any of the following criteria at the time of the baseline visit are NOT eligible to be enrolled in this study:

* Previous Heller myotomy or POEM procedure
* contra-indication to general anesthesia
* Previous mediastinal surgery hiatal hernia greater than 2 cm
* Any anatomical esophageal anomaly that in the opinion of the investigator may render the intervention more difficult, such as sigmoid esophagus on the pre-operative barium swallow or hiatal hernia > 2cm.
* Any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
percent of patients leaving on post-operative day 0 | 1 year

SECONDARY OUTCOMES:
percent of patients who experience post-operative reflux | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Shiwaku H, Inoue H, Sasaki T, Yamashita K, Ohmiya T, Takeno S, Nimura S, Yamashita Y. A prospective analysis of GERD after POEM on anterior myotomy. Surg Endosc. 2016 Jun;30(6):2496-504. doi: 10.1007/s00464-015-4507-0. Epub 2015 Sep 28. PMID 26416381
- [Background] Barbieri LA, Hassan C, Rosati R, Romario UF, Correale L, Repici A. Systematic review and meta-analysis: Efficacy and safety of POEM for achalasia. United European Gastroenterol J. 2015 Aug;3(4):325-34. doi: 10.1177/2050640615581732. PMID 26279840
- [Background] Inoue H, Sato H, Ikeda H, Onimaru M, Sato C, Minami H, Yokomichi H, Kobayashi Y, Grimes KL, Kudo SE. Per-Oral Endoscopic Myotomy: A Series of 500 Patients. J Am Coll Surg. 2015 Aug;221(2):256-64. doi: 10.1016/j.jamcollsurg.2015.03.057. Epub 2015 Apr 11. PMID 26206634
- [Background] Stavropoulos SN, Modayil R, Friedel D. Per oral endoscopic myotomy for the treatment of achalasia. Curr Opin Gastroenterol. 2015 Sep;31(5):430-40. doi: 10.1097/MOG.0000000000000206. PMID 26200001
- [Background] Patel K, Abbassi-Ghadi N, Markar S, Kumar S, Jethwa P, Zaninotto G. Peroral endoscopic myotomy for the treatment of esophageal achalasia: systematic review and pooled analysis. Dis Esophagus. 2016 Oct;29(7):807-819. doi: 10.1111/dote.12387. Epub 2015 Jul 14. PMID 26175119